CLINICAL TRIAL: NCT07203716
Title: Effect of Home-Based and Immediate Pre-Scan Virtual Reality Orientation on Motion Artifacts and Sedation Need in Pediatric MRI: A Three-Arm Randomized Controlled Trial
Brief Title: Preparing Kids for MRI Using VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berker Okay, MD - Pediatrician (Principal Investigator), Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 176-2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Sedation; Child; Virtual Reality; MRI
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental - Home+Booster VR (Experimental): Home exposure 24-48 h pre-scan plus a brief on-site booster immediately before positioning.
  Interventions: Behavioral: Virtual Reality Orientation (Home+Booster)
- Pre-Scan VR Only (Experimental): Single on-site VR exposure immediately before positioning.
  Interventions: Behavioral: Virtual Reality Orientation (Pre-Scan Only)
- Usual Care (Active Comparator): Standard pediatric MRI preparation without VR.
  Interventions: Other: Usual Care (No VR)

INTERVENTIONS:
Behavioral: Virtual Reality Orientation (Home+Booster) — Age-appropriate 360° VR module (~8-10 min) showing MRI room, sounds, positioning, and the importance of keeping still; viewed at home 24-48 h pre-scan on a smartphone/VR viewer (or flat 360° if no headset), plus a brief booster view on site immediately before positioning (~3-5 min refresher).
  Arms: Experimental - Home+Booster VR
Behavioral: Virtual Reality Orientation (Pre-Scan Only) — The same 360° VR module (~8-10 min) viewed once on site in the MRI area immediately before positioning; no home exposure.
  Arms: Pre-Scan VR Only
Other: Usual Care (No VR) — Standard institutional pediatric MRI preparation (verbal explanation, hearing protection demo, child-friendly coaching) without VR.
  Arms: Usual Care

SUMMARY:
Children frequently exhibit pre-MRI anxiety that can cause motion, repeated sequences, prolonged room time, and exposure to sedation. Orientation with Virtual Reality (VR) may reduce anxiety by familiarizing children with the scanner environment and expected sensations. This single-center, three-arm randomized clinical trial evaluates whether (1) Home+Booster VR (an age-appropriate 360° VR module at home ~24-48 hours before MRI plus a brief on-site refresher immediately before positioning), (2) Pre-Scan VR only (same module viewed on site immediately before positioning), or (3) Usual Care without VR improves MRI image quality and tolerance in children undergoing their first-ever MRI.

Eligible participants are children scheduled for clinically indicated, non-emergent MRI with no prior MRI experience. Major exclusions comprise MRI contraindications; contraindications to VR use (e.g., uncontrolled epilepsy or severe motion sickness); uncorrected severe visual/hearing impairment precluding VR viewing; and inability to provide assent/consent. After consent/assent, participants are randomized 1:1:1 to one of three arms. Anticipated enrollment is ~150 total (~50 per arm; up to 60 per arm if feasible). All arms receive routine safety procedures and child-oriented coaching per institutional practice. The VR module (~8-10 minutes) provides a 360° walkthrough of the MRI process (sounds, positioning, keeping still) with child-focused narration. Adherence (timestamps/duration) is recorded where applicable.

The primary outcome is motion artifact rated on a predefined ordinal scale by a board-certified radiologist masked to allocation; the proportion achieving diagnostic quality without repeat/sedation is also reported. Key secondary outcomes include sedation requirement, number of repeated sequences, total scan room time, scan completion without interruption, and change in child anxiety (mYPAS-SF). Additional prespecified measures include comfort/calmness Likert scales, Wong-Baker FACES pain, CEMS during scan, parent state anxiety, satisfaction VAS, physiologic vitals (heart rate, blood pressure, SpO₂) at defined peri-scan time points, observed crying and movement durations, and total scan duration. The trial uses parallel assignment with allocation concealment and masked outcome assessment. Analyses follow intention-to-treat with prespecified subgroup exploration by age bands (5-7 vs 8-10). Recruitment is planned for October 6, 2025; primary completion is expected within approximately three months.

DETAILED DESCRIPTION:
Rationale. Pre-procedural anxiety in pediatric MRI is a well-recognized driver of motion, repetition of sequences, longer scanner occupancy, and sedation exposure. Brief, developmentally tailored exposure using a 360° VR module is hypothesized to reduce anxiety and movement through familiarization with scanner sounds, spatial constraints, and behavioral expectations.

Design Overview. Single-center, three-arm randomized clinical trial with parallel assignment and allocation concealment. Participants with no prior MRI experience are randomized 1:1:1 to Home+Booster VR, Pre-Scan VR only, or Usual Care. Outcome assessment is masked to allocation. Analyses follow intention-to-treat; per-protocol summaries are planned as supportive.

Intervention Content and Delivery. The VR module (~8-10 minutes) depicts arrival, positioning, acoustic noise, and the importance of remaining still. Narration and visuals are age-appropriate.

* Home+Booster VR: module viewed at home approximately 24-48 hours before MRI (re-view permitted), plus a brief on-site refresher immediately before positioning.
* Pre-Scan VR only: module viewed only on site immediately before positioning.
* Usual Care: standard institutional preparation without VR. Routine safety procedures and child-oriented coaching are applied uniformly across arms.

Adherence and Fidelity. Where available, platform logs capture timestamps and duration of module exposure (home and on-site). Staff document completion of on-site viewing and any technical issues. Periodic fidelity checks ensure consistent delivery.

Randomization, Masking, and Allocation Concealment. Randomization is performed via a concealed sequence (computer-generated permuted blocks). Allocation is revealed to staff immediately prior to preparation. Image-quality ratings are performed by a board-certified radiologist masked to allocation. Staff involved in VR delivery are not masked; contact with the assessor is minimized.

Safety Monitoring. VR is paused or discontinued for nausea, dizziness, or discomfort. Standard MRI safety screening is conducted per institutional policy. Adverse events related to VR exposure or MRI are recorded and reviewed by the study team; serious events are reported per institutional requirements.

Data Handling. Data are captured in secure, access-controlled case report forms with predefined range checks. Personally identifiable information is stored separately from analytic datasets. Quality control includes double-entry checks for a subset and automated logic checks.

Statistical Approach (brief). Descriptive statistics summarize baseline characteristics and feasibility metrics (e.g., adherence to the module). The primary endpoint (motion artifact score) is analyzed under intention-to-treat using appropriate ordinal or dichotomous models specified in the statistical analysis plan. Prespecified subgroup analyses examine age bands (5-7 vs 8-10). Multiplicity control procedures are detailed in the analysis plan. Missing data strategies are predefined and documented.

Timeline. Recruitment is planned to commence October 6, 2025. Enrollment and follow-up are expected to conclude within approximately three months, subject to scheduling logistics and scanner availability.

ELIGIBILITY:
Inclusion Criteria:

* Children 5 to 10 years old (inclusive).
* First-ever MRI for a clinically indicated, non-emergent examination (outpatient or elective inpatient).
* Ability to view the age-appropriate 360° VR module (head-mounted viewer or flat 360° on screen) with basic comprehension of instructions (child and/or caregiver in Turkish).
* Parental/guardian informed consent and child assent per age/competence.
* Standard MRI safety screening passed; institutional rescue sedation policies remain available if clinically required.

Exclusion Criteria:

* MRI contraindications (e.g., non-MR-conditional implants, unsafe metallic foreign bodies).
* Pre-planned sedation or general anesthesia irrespective of behavior (clinician decision made prior to randomization).
* Conditions contraindicating VR exposure (e.g., uncontrolled epilepsy, severe motion sickness/vertigo causing intolerance).
* Severe uncorrected visual or hearing impairment precluding module viewing or instruction adherence.
* Emergent/urgent MRI where study procedures could delay care.
* Neurodevelopmental or behavioral conditions that render still positioning entirely unfeasible despite standard coaching (investigator judgment).
* Prior participation in this trial (no re-enrollment).

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Radiologist-Rated MRI Motion Artifact (ordinal score) | During MRI session; assessment completed within 24 hours of image acquisition.
  Motion artifact rated on a pre-specified 4-point ordinal scale per exam by a board-certified radiologist masked to allocation (0 = none; 1 = mild/not affecting diagnostic utility; 2 = moderate/partially limiting; 3 = severe/non-diagnostic). Inter-rater agreement (if applicable) will be summarized separately.
  Unit of Measure: score (0-3)

SECONDARY OUTCOMES:
Diagnostic-Quality MRI Without Repeat or Sedation (yes/no) | At completion of MRI session; determination recorded within 24 hours of image acquisition.
  Proportion of exams achieving diagnostic-quality images without repeated sequences and without sedation, based on pre-specified radiology/report criteria; ratings performed masked to allocation.
  Unit of Measure: percent (%)
Total Scan Room Time | During MRI session (room entry to room exit).
  Time from room entry to room exit during the MRI session, including positioning and image acquisition.
  Unit of Measure: minutes

REFERENCES:
- [Background] van Spaendonck Z, Leeuwenburgh KP, Dremmen M, van Schuppen J, Starreveld D, Dierckx B, Legerstee JS. Comparing Smartphone Virtual Reality Exposure Preparation to Care as Usual in Children Aged 6 to 14 Years Undergoing Magnetic Resonance Imaging: Protocol for a Multicenter, Observer-Blinded, Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 24;12:e41080. doi: 10.2196/41080. PMID 36692931
- [Background] Harned RK 2nd, Strain JD. MRI-compatible audio/visual system: impact on pediatric sedation. Pediatr Radiol. 2001 Apr;31(4):247-50. doi: 10.1007/s002470100426. PMID 11321741
- [Background] Le May S, Genest C, Hung N, Francoeur M, Guingo E, Paquette J, Fortin O, Guay S. The Efficacy of Virtual Reality Game Preparation for Children Scheduled for Magnetic Resonance Imaging Procedures (IMAGINE): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Jun 13;11(6):e30616. doi: 10.2196/30616. PMID 35700000
- [Background] Stunden C, Stratton K, Zakani S, Jacob J. Comparing a Virtual Reality-Based Simulation App (VR-MRI) With a Standard Preparatory Manual and Child Life Program for Improving Success and Reducing Anxiety During Pediatric Medical Imaging: Randomized Clinical Trial. J Med Internet Res. 2021 Sep 22;23(9):e22942. doi: 10.2196/22942. PMID 34550072
- [Background] Ashmore J, Di Pietro J, Williams K, Stokes E, Symons A, Smith M, Clegg L, McGrath C. A Free Virtual Reality Experience to Prepare Pediatric Patients for Magnetic Resonance Imaging: Cross-Sectional Questionnaire Study. JMIR Pediatr Parent. 2019 Apr 18;2(1):e11684. doi: 10.2196/11684. PMID 31518319